CLINICAL TRIAL: NCT01778829
Title: Nasal Intermittent Mandatory Ventilation Versus Continuous Positive Airway Pressure After Extubation of Very Low Birth Weight Infants of the NEOCOSUR Network.
Brief Title: Non Invasive Ventilation Versus Continuous Positive Airway Pressure After Extubation of Very Low Birth Weight Infants.
Acronym: VNINS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Alberto Estay, MD, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sa10i20033
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Neonatal Respiratory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP ventilation mode (Active Comparator): Once the patient is extubated, CPAP ventilation mode is inmediately administered in order to prevent reintubation
  Interventions: Procedure: CPAP ventilation mode
- NIPPV ventilation mode (Experimental): NIPPV: Non Invasive Ventilation mode is administered inmediately after extubation to prevent reintubation
  Interventions: Procedure: NIPPV ventilation mode

INTERVENTIONS:
Procedure: CPAP ventilation mode — Patients are ventilated through a nasal prong coneected to a ventilator that provides a continuous positive airway pressure
  Arms: CPAP ventilation mode
Procedure: NIPPV ventilation mode — Patients are ventilated through a nasal prong connected to a ventilator that provides a non synchronized intermittent positive pressure ventilation
  Arms: NIPPV ventilation mode

SUMMARY:
The purpose of this study is to determine whether Nasal intermittent positive pressure ventilation (NIPPV) non synchronized is better than continuous positive airway pressure (NCPAP)in preventing extubation failure within 72 h, after extubation of very low birth weight infants at the NEOCOSUR Network.

DETAILED DESCRIPTION:
Is a Randomized trial to preterms infants <1500g and less than 34 weeks with RDS requiring machanical ventilation in the extubation period, randomized to receive NIPPV or NCPAP once extubation criteria were met. Parental written informed consent is required previous extubation. The failure rate is defined as the need for re-intubation and mechanical ventilation).

Exclusion criteria are: major congenital anomalies; presence of cardiovascular instability;intubation less than 2 hours; mechanical ventilation more than 14 days, using muscle relaxant, airway anomalies, consent not provided or refused.

Outcome measures:

The primary outcome was to assess the need for re-intubation within the first 72 hours after extubation in the 2 groups.

The criteria for failure were met by at least 1 of the following:

pH < 7.25 and PaCO2 > 65 mmHg; recurrent apnea more than 2 episodes per hour associated with bradycardia; during 4 hour continuous; 2 episodes of apnea that required bagand-mask ventilation in any time during the study; or a PaO2 < 50 mm Hg with a fraction of inspired oxygen > 0.6. The secondary outcomes concerning respiratory support were total duration on ETT ventilation, total duration on NCPAP, total duration on supplemental oxygen, incidence of pneumothorax,BPD and dead. Other outcomes included incidence of patent ductus arteriosus (PDA), necrotizing enterocolitis, intraventricular hemorrhage grades 3 and 4, retinopathy of prematurity stage 3, time to full feeds, and length of hospital stay.

Sample size calculations for the primary outcome: We estimated that there would be a more than 80% chance of detecting 43% difference between the groups (alpha 0.05) when samplesize (n) is 110 patients for each mode of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Preterm with a weight less than 1501 g
* Gestational age less or equal to 34 weeks
* Preterm that meets extubation criteria after at least 2 hours and less than 14 days connected to mechanical ventilation
* Patient receiving methylxanthynes

Exclusion Criteria:

* Patient more than 14 days in mechanical ventilation
* Newborn with congenital cardiopathy
* Newborn with congenital malformation
* Newborn wirh chromosomopathy or genopathic disease
* Newborn with suspected gastrointestinal disease
* Newborn with neuromuscular disease or receiving muscle relaxants
* Lack or informed consent signed by parents or legal representative

Ages: 2 Hours to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | apnea rate and respiratory failure.
  The criteria for failure were met by at least 1 of the following:
  pH less than 7.25 and PaCO2 over 65 mmHg; recurrent apnea more than 2 episodes per hour associated with bradycardia; during 4 hour continuous; 2 episodes of apnea that required bagand-mask ventilation in any time during the study; or a PaO2 less than 50 mm Hg with a fraction of inspired oxygen over 0.6.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Estay, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clinico, Pontificia Universidad Catolica de Chile, Santiago, Chile

REFERENCES:
- [Derived] Estay AS, Mariani GL, Alvarez CA, Milet B, Agost D, Avila CP, Roldan L, Abdala DA, Keller R, Galletti MF, Gonzalez A; for the NEOCOSUR Neonatal Network. Randomized Controlled Trial of Nonsynchronized Nasal Intermittent Positive Pressure Ventilation versus Nasal CPAP after Extubation of VLBW Infants. Neonatology. 2020;117(2):193-199. doi: 10.1159/000506164. Epub 2020 May 8. PMID 32388511